CLINICAL TRIAL: NCT04037969
Title: Comparison of Tear Evaporation Rate With DAILIES TOTAL1 and Biotrue ONEday
Acronym: MALTESE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 41195
Record Dates: First submitted 2019-07-26; First posted 2019-07-30 (Actual); Results first posted 2021-04-23 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-03

CONDITIONS: Evaporative Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants and investigators are masked as to which lens is assigned to each eye.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Nesofilcon A/Delefilcon A (Experimental): Nesofilcon A was worn in right eye and delefilcon A worn in the left eye.
  Interventions: Device: Nesofilcon A; Device: Delefilcon A
- Delefilcon A/Nesofilcon A (Experimental): Delefilcon A was worn in right eye and Nesofilcon A worn in the left eye.
  Interventions: Device: Nesofilcon A; Device: Delefilcon A

INTERVENTIONS:
Device: Nesofilcon A — Hydrogel contact lens for daily wear
Device: Delefilcon A — Silicone hydrogel contact lens for daily wear

SUMMARY:
The purpose of this pilot study is to compare the effect of DAILIES TOTAL1, a low water content silicone hydrogel lens, and Biotrue ONEday, a high water content hydrogel lens, on the rate of tear evaporation. The study will also serve to validate the novel, in-house developed evaporimeter.

ELIGIBILITY:
Inclusion Criteria:

1. Is at least 17 years of age and has full legal capacity to volunteer;
2. Has read and signed an information consent letter;
3. Is willing and able to follow instructions and maintain the appointment schedule;
4. Has worn soft contact lenses for a minimum of 6 months;
5. Currently wears soft contact lenses for at least 4 days per week and 8 hours per day;
6. Has an acceptable fit and comfort with both study contact lenses in the powers available;
7. Has less than or equal to 1.00DS difference between eyes in their habitual contact lenses;
8. Is willing to be awake for at least 2 hours before visit 2;
9. Is willing to not wear eye makeup on the day of visit 2 and 3;
10. Is willing to not use eye drops or artificial tears on the day of visits 1, 2, and 3;
11. Has a wearable pair of spectacles.

Exclusion Criteria:

1. Is participating in any concurrent clinical or research study;
2. Has any known active* ocular disease and/or infection;
3. Has a systemic condition that in the opinion of the investigator may affect a study outcome variable;
4. Is using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable;
5. Has known sensitivity to sodium fluorescein dye;
6. Is pregnant, lactating or planning a pregnancy at the time of enrolment (by verbal confirmation at the screening visit);
7. Is aphakic;
8. Has undergone refractive error surgery;
9. Has a known sensitivity to petroleum jelly (Vaseline);
10. Has epilepsy and/or a sensitivity to flashing lights;
11. Wears toric contact lenses;
12. Has any physical impairment that would interfere with holding the evaporimeter;
13. Has taken part in another research study within the last 14 days.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-08-07 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2019-11-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Ocular Research & Education, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Nesofilcon A/Delefilcon A: Nesofilcon A randomly assigned to one eye with delefilcon A in the fellow eye.
  Nesofilcon A: Hydrogel contact lens for daily wear
- Delefilcon A/Nesofilcon A: Delefilcon A randomly assigned to one eye with nesofilcon A in the fellow eye.
  Delefilcon A: Silicone hydrogel contact lens for daily wear
Period: Overall Study
Arm/Group | Nesofilcon A/Delefilcon A | Delefilcon A/Nesofilcon A
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nesofilcon A/Delefilcon A | Delefilcon A/Nesofilcon A | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 10 | 19
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.2 (17.1) | 25.1 (9.6) | 28.2 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 1 | 0 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Tear Evaporation Rate With Nesofilcon A
Description: Tear film evaporation rate (% relative humidity per second) was performed using a novel evaporimeter as a non-invasive measurement of tear film evaporation. The slope was calculated from the change in humidity between 7 to 17.5 seconds while the eye was open and between 10 to 17.5 seconds when the eye was closed. Data from the both eyes were analyzed.
Time Frame: Baseline, 15 minutes post-contact lens, 6 hours post-contact lens
Measure: Mean (Standard Deviation); unit: % relative humidity per second
Groups:
- Full Group: Delefilcon A was worn in a randomly assigned eye and Nesofilcon A was worn in the fellow eye.
  Nesofilcon A: Hydrogel contact lens for daily wear
  Delefilcon A: Silicone hydrogel contact lens for daily wear
Arm/Group | Full Group
Number analyzed (Participants) | 20
% relative humidity per second
  Baseline | 0.81 (0.30)
  15 minutes post-contact lenses | 0.88 (0.32)
  6 hours post-contact lenses | 0.92 (0.38)

2. Primary Outcome: Tear Evaporation Rate With Delefilcon A
Description: as for outcome 1
Time Frame: Baseline, 15 minutes post-contact lens, 6 hours post-contact lens
Measure: Mean (Standard Deviation); unit: % relative humidity per second
Arm/Group | Full Group
Number analyzed (Participants) | 20
% relative humidity per second
  Baseline | 0.74 (0.21)
  15 minutes post-contact lenses | 0.87 (0.24)
  6 hours post-contact lenses | 0.95 (0.30)

ADVERSE EVENTS:
Time Frame: One day
Arm/Group | Nesofilcon A/Delefilcon A | Delefilcon A/Nesofilcon A
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-24): https://cdn.clinicaltrials.gov/large-docs/69/NCT04037969/Prot_SAP_000.pdf